CLINICAL TRIAL: NCT03596658
Title: Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of SHR9549 in Women With ER Positive HER2 Negative Advanced Breast Cancer
Brief Title: SHR9549 in ER Positive HER2 Negative Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR9549-I-101
Record Dates: First submitted 2018-06-25; First posted 2018-07-24 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2018-07

CONDITIONS: ER+ HER2- Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR9549 dose escalation and expansion(s) (Experimental): Escalating dose of SHR9549 with intensive safety monitoring to ensure the safety of patients
  Interventions: Drug: SHR9549

INTERVENTIONS:
Drug: SHR9549 — If initial dosing of SHR9549 is tolerated then subsequent cohorts will test increasing doses until a maximum tolerated dose(MTD) is defined
  Other Names: SHR9549 tablet

SUMMARY:
This is a phase 1 open label multicentre study of SHR9549 administered orally in patients with advanced estrogen receptor (ER) positive human epidermal receptor 2 (HER2) negative breast cancer. The study design allows an escalation of dose with intensive safety monitoring to ensure the safety of patients. The study will determine the maximum tolerated dose(MTD). In addition, expansion cohort(s) at potential therapeutic dose(s) in patients will be enrolled to further determine the safety, tolerability, pharmacokinetics and biological activity of SHR9549.

DETAILED DESCRIPTION:
A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of SHR9549 in Women with Estrogen Receptor (ER) Positive Human Epidermal Receptor (HER-2) Negative Advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years.
* Confirmation of ER positive; HER2 negative Advanced breast cancer
* Documented disease progression after at least 6 months prior endocrine therapy for ER positive breast cancer.
* Receipt of ≤2 lines of prior chemotherapy for advanced disease.
* Any menopausal status.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 and with minimum life expectancy of 12 weeks.

Exclusion Criteria:

* Any anti-cancer drugs for the treatment of advanced breast cancer within 14 days of the first dose of study treatment.
* Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment with the exception of alopecia.
* Patient who is unsuitable for endocrine therapy alone including presence of life-threatening metastatic visceral disease.
* uncontrolled central nervous system metastatic disease.
* Any evidence of severe or uncontrolled systemic diseases.
* Inadequate bone marrow reserve or organ function.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | baseline through 28 days
  to determine DLT in order to assess the tolerability of SHR9549
Maximum Tolerated Dose (MTD) | baseline through 28 days
  to determine MTD in order to assess the tolerability of SHR9549

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | baseline through 12 weeks
  Single and multiple dose pharmacokinetic parameters of SHR9549 at pre-defined intervals
Area under the plasma concentration versus time curve (AUC) | baseline through 12 weeks
  Single and multiple dose pharmacokinetic parameters of SHR9549 at pre-defined intervals
overall response rate (ORR) | every 8 weeks for 24 weeks and then every 12 weeks thereafter through study completion, an average of 6 months
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
progression free survival (PFS) | every 8 weeks for 24 weeks and then every 12 weeks thereafter through study completion, an average of 6 months
  Antitumour activity evaluation by following up patients' progression and survival
Incidence of Treatment-Emergent Adverse Events | baseline through 30 days after study completion
  to assess the safety of SHR9549

CONTACTS AND LOCATIONS:
Locations (1):
- The 307th Hospital of Military Chinese People's Liberation Army, Beijing, Beijing Municipality, China